CLINICAL TRIAL: NCT01432444
Title: Open-label Study to Assess Hospitalization Rates in Adult Schizophrenic Patients Treated With Oral Antipsychotics for 6 Months and IM Depot Aripiprazole for 6 Months, Respectively, in a Naturalistic Community Setting
Brief Title: Open-label Study to Compare Hospitalization Rates of Schizophrenic Patients Treated With Oral Antipsychotics Versus IM Depot Aripiprazole
Acronym: ARRIVE US
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-11-283
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-14597 (Experimental): Aripiprazole IM depot injection 300 mg or 400 mg.
  Interventions: Drug: Aripiprazole (Abilify®) IM Depot Injection

INTERVENTIONS:
Drug: Aripiprazole (Abilify®) IM Depot Injection — 400 mg IM depot injection every 26-30 days. Dosage may be adjusted at the investigator's discretion to 300 mg.
  Number of injections: 6. Subjects have the option of entering the extension phase of the study and continuing with injections every 26-30 days until the drug is either commercially available, or December 2013.
  Other Names: ABILIFY®

SUMMARY:
The purpose of this study is to compare retrospective hospitalization rates of schizophrenic patients treated with oral antipsychotics to prospective hospitalization rates of these patients treated with IM depot aripiprazole.

DETAILED DESCRIPTION:
Nonadherence to antipsychotic medications remains a frequent cause of relapse among patients with schizophrenia, increasing hospitalization rates, hospitalization days, and hospitalization costs. Among hospitalized adults, schizophrenia is the fourth most commonly diagnosed illness and has the seventh longest mean duration of hospital stay in the US. Frequent relapses and hospitalization can affect quality of life in these patients. Long-acting injections (intramuscular depot) antipsychotic medication is a means to treatment adherence and increased quality of life for patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to provide written informed consent. If the IRB requires consent by a legally acceptable representative in addition to the subject, all required consents must be obtained prior to any protocol-required procedure.
* Male and female subjects 18 to 65 years of age, inclusive.
* Current diagnosis of schizophrenia as defined by DSM-IV-TR criteria and a history of the illness for at least 1 year (12 months).
* Subjects who in the investigator's judgment would benefit from extended treatment with a long-acting injectable formulation.
* Subjects who have at least 1 inpatient psychiatric hospitalization in the 4 years (48 months) prior to screening, but have been managed as outpatients for the 4 weeks prior entering the study.
* Subjects must have been on oral antipsychotic treatment for the full 7 months prior to the screening phase.
* Subjects who have shown response to previous antipsychotic treatment.
* Subjects who understand the nature of the trial and are able to follow the protocol requirements.

Exclusion Criteria:

* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated), or have been incarcerated in the past 7 months for any reason must not be enrolled into this trial.
* Subjects who may require potent CYP2D6 or CYP3A4 inhibitors or CYP3A4 inducers during the trial.
* Any subject who requires or may need any other antipsychotic medications during the course of the trial, other than allowed rescue medication.
* Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones.
* Subjects with a history of hypersensitivity to antipsychotic agents.
* Subjects deemed intolerant of receiving injectable treatment.
* Subjects who have received electroconvulsive therapy within the last 7 months prior to screening.
* Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia as assessed by the investigator.
* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Subjects requiring hospitalization for any psychiatric reason during the 4 weeks prior to signing the ICF or during the screening period.
* Subjects without at least 1 inpatient psychiatric hospitalization in the last 4 years (48 months) prior to screening.
* Subjects who have met DSM-IV-TR criteria for any significant substance use disorder within 3 months prior to screening.
* Subjects who are considered treatment-resistant to antipsychotic medication other than clozapine.
* Treatment with long-acting injectable antipsychotics in which the last dose was within 7 months prior to screening.
* Subjects who have not been treated with oral antipsychotics for 7 months prior to screening.
* Subjects who have a significant risk of committing suicide
* Subjects who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial.
* Females who are pregnant or lactating, sexually active males and females who will not commit to utilizing birth control during the trial and for up to 180 days following the trial.
* Abnormal laboratory or physical examination results indicating a condition which may interfere with the results of the study or pose a safety risk to the subject.
* Subjects who have previously enrolled in an aripiprazole IM depot clinical study, except for subjects entering this trial from the Canadian 31-11-284 trial.
* Subjects who have participated in any clinical trial with an investigational agent within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cox, MD, Study Director — Kevin.TC-Cox@otsuka-us.com
Locations (105):
- United States (100):
  - Dothan, Alabama
  - Tucson, Arizona
  - Fayetteville, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Bellflower, California
  - Carson, California
  - Costa Mesa, California
  - Downey, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Los Angeles, California
  - National City, California
  - Norwalk, California
  - Oakland, California
  - Oceanside, California
  - Orange, California
  - Palo Alto, California
  - Paramount, California
  - Pasadena, California
  - Riverside, California
  - San Diego, California
  - San Francisco, California
  - Santa Ana, California
  - Torrance, California
  - Middletown, Connecticut
  - New Brittain, Connecticut
  - Norwalk, Connecticut
  - Boynton Beach, Florida
  - Coral Gables, Florida
  - Doral, Florida
  - Hialeah, Florida
  - Jacksonville Beach, Florida
  - Miami, Florida
  - Oakland Park, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Saint Augustine, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Joliet, Illinois
  - Naperville, Illinois
  - South Bend, Indiana
  - Topeka, Kansas
  - Witchita, Kansas
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Newton, Massachusetts
  - Bloomfield Hills, Michigan
  - Grand Rapids, Michigan
  - Paw Paw, Michigan
  - Minneapolis, Minnesota
  - Creve Coeur, Missouri
  - Kansas City, Missouri
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - North Platte, Nebraska
  - Sparks, Nevada
  - Nashua, New Hampshire
  - Albuquerque, New Mexico
  - Amherst, New York
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Wards Island, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Canton, Ohio
  - Centennial, Ohio
  - Garfield Heights, Ohio
  - Mason, Ohio
  - Oklahoma City, Oklahoma
  - McMurray, Pennsylvania
  - Phoenixville, Pennsylvania
  - Scranton, Pennsylvania
  - Sellersville, Pennsylvania
  - Sioux Falls, South Dakota
  - Franklin, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Wharton, Texas
  - Salt Lake City, Utah
  - Bellevue, Washington
  - Bothell, Washington
  - Kirkland, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Canada (5):
  - Penticton, British Columbia
  - Halifax, Nova Scotia
  - Brampton, Ontario
  - Chatham, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Peters-Strickland T, Zhao C, Perry PP, Eramo A, Salzman PM, McQuade RD, Johnson BR, Sanchez R. Effects of aripiprazole once-monthly on symptoms of schizophrenia in patients switched from oral antipsychotics. CNS Spectr. 2016 Dec;21(6):460-465. doi: 10.1017/S1092852916000365. Epub 2016 Aug 17. PMID 27531181
- [Derived] Kane JM, Zhao C, Johnson BR, Baker RA, Eramo A, McQuade RD, Duca AR, Sanchez R, Peters-Strickland T. Hospitalization rates in patients switched from oral anti-psychotics to aripiprazole once-monthly: final efficacy analysis. J Med Econ. 2015 Feb;18(2):145-54. doi: 10.3111/13696998.2014.979936. Epub 2014 Nov 10. PMID 25347448
- [Derived] Kane JM, Sanchez R, Zhao J, Duca AR, Johnson BR, McQuade RD, Eramo A, Baker RA, Peters-Strickland T. Hospitalisation rates in patients switched from oral anti-psychotics to aripiprazole once-monthly for the management of schizophrenia. J Med Econ. 2013 Jul;16(7):917-25. doi: 10.3111/13696998.2013.804411. Epub 2013 May 28. PMID 23663091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study assessed hospitalization rates in adults with schizophrenia treated prospectively for 6 months with aripiprazole intramuscular depot compared with 6 month retrospective treatment with oral antipsychotics. The study comprised 3 phases: Tolerability/Cross-titration (Phase A), Open-label Aripiprazole (Phase B), Extension (Phase C).
Pre-assignment Details: 493 participants were enrolled, 325 of which had no history of tolerating oral aripiprazole entered Phase A, all participants completed Phase A combined with remainder of participants to enter Phase B. All outcome measures were assessed in Phase B.
Groups:
- Tolerability/Cross-titration Phase (Phase A): In Phase A, participants who had no history of tolerating oral aripiprazole entered a Tolerability Assessment/Cross-titration Phase in order to assess tolerability to oral aripiprazole. The recommended initial dose of oral aripiprazole in the Tolerability Assessment/Cross-titration Phase was 10 mg or 15 mg/day, depending on the participant's symptoms and the study physician's judgment. Participants were seen in the clinic at baseline and weekly thereafter for a minimum of 1 week and maximum of 4 weeks/28 days, until tolerability to oral aripiprazole had been determined, based on physician's discretion, or until the participant was terminated from the study.
- Open-label Aripiprazole IM Depot Treatment Phase (Phase B): In Phase B, all participants received aripiprazole IM depot 400 mg and had received supplemental oral aripiprazole for the first 14 days of Phase B (open-label aripiprazole IM depot treatment phase) for more than or equal to 3 months. However, at the discretion of the study physician, the dose of aripiprazole IM depot was decreased to 300 mg only if needed for tolerability and subsequently increased the dose to 400 mg for efficacy as required. This dose adjustment was permitted as often as necessary to maintain symptomatic stability with acceptable tolerability. For purposes of this study, participants who completed Week 24 of Phase B were defined as trial completers.
- Extension Phase (Phase C): Participants who completed the 24-Week treatment period (Phase B), and whom the study physician believes would receive benefit from continued treatment with aripiprazole IM depot, were eligible to enter Phase C. During Phase C, participants were to continue treatment with aripiprazole IM depot until approximately 400 subjects have enrolled in Phase B (in order to achieve approximately 200 Phase B completers).
Period: Tolerability/Cross-titration Phase
Arm/Group | Tolerability/Cross-titration Phase (Phase A) | Open-label Aripiprazole IM Depot Treatment Phase (Phase B) | Extension Phase (Phase C)
Started | 325 | 0 | 0
Completed | 265 | 0 | 0
Not Completed | 60 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0
Not completed — Adverse Event | 16 | 0 | 0
Not completed — Met Withdrawal Criteria | 5 | 0 | 0
Not completed — Physician Decision | 8 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0
Period: Treatment Phase
Arm/Group | Tolerability/Cross-titration Phase (Phase A) | Open-label Aripiprazole IM Depot Treatment Phase (Phase B) | Extension Phase (Phase C)
Started | 0 | 433 | 0
Completed | 0 | 293 | 0
Not Completed | 0 | 140 | 0
Not completed — Lost to Follow-up | 0 | 33 | 0
Not completed — Adverse Event | 0 | 37 | 0
Not completed — Met Withdrawal Criteria | 0 | 11 | 0
Not completed — Physician Decision | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 41 | 0
Not completed — Protocol Deviation | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 10 | 0
Period: Extension Phase
Arm/Group | Tolerability/Cross-titration Phase (Phase A) | Open-label Aripiprazole IM Depot Treatment Phase (Phase B) | Extension Phase (Phase C)
Started | 0 | 0 | 192
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 192
Not completed — Lost to Follow-up | 0 | 0 | 17
Not completed — Adverse Event | 0 | 0 | 10
Not completed — Sponsor Discontinued Trial | 0 | 0 | 7
Not completed — Met Withdrawal Criteria | 0 | 0 | 144
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B)
Number analyzed (Participants) | 433
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 301

OUTCOME MEASURES:

1. Primary Outcome: Number of Inpatient Psychiatric Hospitalization for Retrospective Period (Months 4-6) and Prospective Period (Months 4-6).
Description: The comparison of inpatient psychiatric hospitalization rates (proportion of patients with ≥ inpatient psychiatric hospitalizations) between the retrospective period months 4-6 (Weeks-12 to -24) while on oral standard of care antipsychotic treatment and the prospective period Phase B months 4-6 (Weeks 12 to 24) after the switch to aripiprazole IM depot. Open-label Aripiprazole IM Depot Treatment Phase 3-month Completer sample comprised of all participants who entered open-label aripiprazole IM depot treatment Phase and completed at least 3 months of treatment. This sample was used for the primary endpoint analysis (N=336).
Time Frame: Retrospective period Months 4-6; Prospective period Months 4-6
Population: The core dataset for all efficacy analyses is the Intent-to-Treat (ITT) dataset which consisted of data from all participants who entered Phase B regardless of receiving a dose in the Open-label Aripiprazole IM Depot Treatment Phase.
Measure: Number; unit: participants
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B)
Number analyzed (Participants) | 336
participants
  Retrospective period | 91 (0.6)
  Prospective period | 9 (0.2)
Statistical Analysis 1: Comparison: Open-label Aripiprazole IM Depot Treatment Phase (Phase B); Inpatient hospitalization for retrospective period (Months 4-6) and prospective period (Months 4-6) for closed or open unit; Test type: Superiority or Other; p < .0001, McNemar — P-value was derived from Exact McNemar test

2. Secondary Outcome: Change From Baseline in PANSS (Positive and Negative Syndrome Scale) Total Score.
Description: The PANSS consists of three subscales with a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicates (absence of symptoms) and a score of 7 indicates (extremely severe symptoms). The symptom constructs for each subscale are as follows: 7 Positive subscale symptom constructs, 7 Negative subscale symptom constructs and 16 General Psychopathology subscale symptom constructs. The PANSS total score ranges from 30 to 210.
Time Frame: Baseline to Week 24
Population: The core dataset for all efficacy analyses is the ITT dataset which consisted of data from all participants who entered Phase B regardless of receiving a dose in the Open-label Aripiprazole IM Depot Treatment Phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B)
Number analyzed (Participants) | 427
Units on a scale
  Week 4 (N= 390) | -7.9 (14.0)
  Week 12 (N= 410) | -8.4 (15.6)
  Week 24 (N= 410) | -8.4 (17.7)
Statistical Analysis 1: Comparison: Open-label Aripiprazole IM Depot Treatment Phase (Phase B); Statistical analyses for Week 4, 12 and 24; Test type: Superiority or Other; p < .0001, t-test — Derived from T-test of Mean=0; Mean duration was derived as the cumulative duration divided by the number of inpatient non-psychiatric hospitalization

3. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score.
Description: The PANSS consists of three subscales with a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicates (absence of symptoms) and a score of 7 indicates (extremely severe symptoms). The symptom constructs for each subscale are as follows: 7 Positive subscale symptom constructs, 7 Negative subscale symptom constructs and 16 General Psychopathology subscale symptom constructs. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity suspiciousness/ persecution, and hostility. The PANSS Positive Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B)
Number analyzed (Participants) | 427
Units on a scale
  Week 4 (N= 390) | -2.7 (4.4)
  Week 12 (N= 410) | -2.9 (4.9)
  Week 24 (N= 410) | -3.0 (5.4)
Statistical Analysis 1: Comparison: Open-label Aripiprazole IM Depot Treatment Phase (Phase B); Statistical analyses for Week 4, Week 12 and Week 24; Test type: Superiority or Other; p < .0001, t-test, 2 sided — Derived from T-test of Mean=0; Mean duration was derived as the cumulative duration divided by the number of inpatient non-psychiatric hospitalization

4. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score.
Description: The PANSS consists of three subscales with a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicates (absence of symptoms) and a score of 7 indicates (extremely severe symptoms). The symptom constructs for each subscale are as follows: 7 Positive subscale symptom constructs, 7 Negative subscale symptom constructs and 16 General Psychopathology subscale symptom constructs. The 7 negative symptom constructs are blunted affect, emotional withdrawal, poor rapport, passive pathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS Negative Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B)
Number analyzed (Participants) | 427
Units on a scale
  Week 4 | -1.7 (4.6)
  Week 12 | -1.6 (5.1)
  Week 24 | -1.6 (5.8)
Statistical Analysis 1: Comparison: Open-label Aripiprazole IM Depot Treatment Phase (Phase B); Statistical analysis for Week 4, 12 and 24; Test type: Superiority or Other; p < .0001, t-test, 2 sided — Derived from T-test of Mean=0; Mean duration was derived as the cumulative duration divided by the number of inpatient non-psychiatric hospitalization

5. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity Score (CGI-S).
Description: The severity of illness for each participant were rated using the CGI-S scale. To assess CGI-S, study physician were to answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B)
Number analyzed (Participants) | 425
Units on a scale
  Week 4 (N= 391) | -0.3 (0.8)
  Week 12 (N= 410) | -0.4 (0.9)
  Week 24 (N= 410) | -0.5 (1.0)
Statistical Analysis 1: Comparison: Open-label Aripiprazole IM Depot Treatment Phase (Phase B); Statistical analysEs for Week 4, 12 and 24; Test type: Superiority or Other; p < .0001, t-test — Derived from t-test of mean=0

6. Secondary Outcome: Mean Clinical Global Impression-Improvement Score (CGI-I) by Week.
Description: The efficacy of trial medication was rated for each participant using the CGI-I scale. The study physician would rate the participants total improvement whether or not it was entirely due to drug treatment. All responses were compared to the participants condition at Baseline of the appropriate phase. The CGI-I during Phase B were assessed relative to the participants condition at the Phase B Baseline visit. Response choices included: 0 = not assessed; 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Week 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B)
Number analyzed (Participants) | 425
Units on a scale
  Week 4 (N= 283) | 2.9 (0.9)
  Week 12 (N= 293) | 2.7 (1.0)
  Week 24 (N= 293) | 2.5 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from ICF signed until Follow-up 30 (± 3) days after last visit.
Description: 431 participants who had received at least one dose of study medication in the corresponding trial phase were included in the safety analysis.
Groups:
- Extension Phase (Phase C): Participants who completed the 24-Week treatment period (Phase B), and whom the study physician believed would benefit from continued treatment with aripiprazole IM depot, were eligible to enter Phase C. During Phase C, participants were to continue treatment with aripiprazole IM depot until approximately 400 subjects have enrolled in Phase B (in order to achieve approximately 200 Phase B completers).
Arm/Group | Open-label Aripiprazole IM Depot Treatment Phase (Phase B) | Extension Phase (Phase C)
Serious Adverse Events (participants affected / at risk) | 61/431 | 19/192
Other Adverse Events (participants affected / at risk) | 60/431 | 24/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Aripiprazole IM Depot Treatment Phase (Phase B) (N=431) | Extension Phase (Phase C) (N=192)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetis mellitus (Metabolism and nutrition disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 4 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Psychotic disorder (Psychiatric disorders) | 8 | 3
Schizophrenia (Psychiatric disorders) | 11 | 6
Schizophrenia, paranoid type (Psychiatric disorders) | 14 | 3
Schizophrenia, undifferentiated type (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 6 | 1
Suicide attempt (Psychiatric disorders) | 3 | 1
Penile oedema (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Aripiprazole IM Depot Treatment Phase (Phase B) (N=431) | Extension Phase (Phase C) (N=192)
Akathisia (Nervous system disorders) | 27 | 9
Insomnia (Psychiatric disorders) | 29 | 6
Weight increased (Investigations) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No